CLINICAL TRIAL: NCT03171272
Title: Effects of Inspiratory Muscle Training on the Functional Gait Performance of Individuals After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lorena de Oliveira Vaz Miranda (Other)
Responsible Party: Sponsor-Investigator, Lorena de Oliveira Vaz Miranda, Principal Investigator, Graduated in Physiotherapy by UFMG (2009) and specialist in Respiratory Physiotherapy by ASSOBRAFIR (2016), Sarah Network of Rehabilitation Hospitals
Organization: Sarah Network of Rehabilitation Hospitals (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 65028517.0.0000.0022
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Stroke; Inspiratory Muscle Training; Quality of Life; Gait
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Other: Inspiratory Muscle Training
- Control Group (Sham Comparator)
  Interventions: Other: Inspiratory Muscle Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — Experimental: IMT will include training of the inspiratory muscles five times per week over six weeks, divided into two fiftten-minute sessions of inspiratory training totaling 30 minutes of training. Thresholds regulated at 50% of the subjects' maximal inspiratory pressure values, the load being increased weekly. Associated with the IMT, subjects will participate in the rehabilitation program, when they will perform 7 sessions of physiotherapy per week, totaling 42 sessions, as well as 180 minutes per week of aerobic exercise, for six weeks.
  Sham Group: This group will underwent exactly the same protocol but the participants will receive the threshold devices with the minimum resistance of the spring, which will be also concealed. The control group will also participate in the rehabilitation program and undergo the same procedures, except for the load adjustments.

SUMMARY:
The most commonly observed sequel after stroke is muscle weakness, which can also be identified in respiratory muscles, in the acute and chronic phases, and may compromise the lung function of these individuals. Studies have shown that lower Pimax values are found in non-community ambulators, and gait velocity has been reported as an important indicator of functionality after stroke, with higher gait velocity values associated with greater community participation and better quality of life.

This study will test the hypothesis that training of the inspiratory muscles is effective in improving strength and endurance of the inspiratory muscles and functionality, including speed of gait, functional gait perfomarnce, activities of daily living and quality of life with stroke subjects.

For this clinical trial, people after stroke will be randomly allocated into either experimental or control/sham groups. The experimental group will undertake training of the inspiratory muscles with the Power Breath Medical Classic device regulated at 50% of the subjects' maximal inspiratory pressure values, five times/week over six weeks, twice a day for 15 minutes, totaling 30 minutes/day. The control group will undertake the same protocol, but the participants will receive the devices with a minimal load, wich corresponds to 1cmH2O. Both groups will participate in the rehabilitation program for 6 weeks. At baseline and post intervention, after the cessation of the interventions, researchers blinded to group allocations will collect the following outcome measures: maximal respiratory pressures, respiratory muscle endurance, functional gait performance, activities of daily living and quality of life. After 12 weeks will collect again maximal inspiratory pressures and functional gait performance.

DETAILED DESCRIPTION:
The most commonly observed sequel after stroke is muscle weakness, which can also be identified in respiratory muscles, in the acute and chronic phases, and may compromise the lung function of these individuals. Studies have shown that lower Pimax values are found in non-community ambulators, and gait velocity has been reported as an important indicator of functionality after stroke, with higher gait velocity values associated with greater community participation and better Quality of life.

Aim: This study will test the hypothesis that training of the inspiratory muscles is effective in improving strength and endurance of the inspiratory muscles and functional gait perfomarnce, activities of daily living and quality of life with stroke subjects.

Design: For this prospective, triple-blinded, randomized clinical trial, people after stroke will be randomly allocated into either experimental or control/sham groups. The experimental group will undertake training of the inspiratory muscles with the PowerBreath Medic Plus regulated at 50% of the subjects' maximal inspiratory pressure (MIP) values, five times/week over six weeks during 30 minutes/day. The control group will undertake the same protocol, but the participants will receive the threshold devices with minimal resistance valves. At baseline and post intervention after the cessation of the interventions, researchers blinded to group allocations will collect all outcome measures. After 12 weeks will collect again maximal inspiratory pressures and functional gait performance.

Study outcomes: Primary outcomes will be functional gait perfomarnce. Secondary outcomes will include inspiratory endurance, activities of daily living and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adults with hemiparesis after stroke, of any etiology, ischemic or hemorrhagic, that carry out walking with or without assistance locomotion; Aged between 18 and 80 years of age; In the chronic period (between 6 months and 5 years); clinically stable (Measured through clinical and hemodynamic stability: vital signs within normal and released for physical activity by the physician), who present with inspiratory muscle weakness, defined as Pimáx less than -80cmH2O and score in the normal Mini Mental State Examination (MMSE) For schooling.

Exclusion Criteria:

* Smokers and ex-smokers for more than five years, presence of facial paralysis that prevents lip occlusion, associated neurological diseases, orthopedic alterations that include distortions of the chest cavity or pains that prevent the tests from being performed, respiratory dysfunctions, cardiac dysfunctions that Compromise hemodynamic stability.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
change in functional gait perfomarnce | change from Baseline at 6 weeks
  functional gait perfomarnce will be assessed by six minute walk test. (6MWT)

SECONDARY OUTCOMES:
endurance muscular respiratory | Baseline and after 6 weeks
  inspiratory and expiratory endurance will be assessed by the threshold devices, following previously described protocols.
maximal respiratory pressures | Baseline, after 6 six weeks and three-monsth follow-ups
  Maximal respiratory pressures will be assessed by a analogic manovacuometer, following previously described protocols.
functional gait perfomarnce | three-monsth follow-ups
  functional gait perfomarnce will be assessed by six minute walk test. (6MWT)
activities of daily living | Baseline and after 6 weeks
  activities of daily living: will be assessed by measure independence functional (MIF)
Quality of life | Baseline, after 6 weeks and three-monsth follow-ups
  Quality of life will be assessed by the Brazilian version of the EQ5D.

CONTACTS AND LOCATIONS:
Overall Officials: Jamary Oliveira Filho, Study Director — Federal University of Bahia
Locations (1):
- Lorena de Oliveira Vaz Miranda, Salvador, Estado de Bahia, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data collected in this study will be made available on this basis and will be published in a scientific journal. A master's dissertation will also be built. Further said reports will be provided to the ethics committee while conducting the study.

REFERENCES:
- [Derived] Vaz LO, Almeida JC, Froes KSDSO, Dias C, Pinto EB, Oliveira-Filho J. Effects of inspiratory muscle training on walking capacity of individuals after stroke: A double-blind randomized trial. Clin Rehabil. 2021 Sep;35(9):1247-1256. doi: 10.1177/0269215521999591. Epub 2021 Mar 11. PMID 33706569